CLINICAL TRIAL: NCT06020014
Title: A Phase 2a Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of AZD4604 Twice Daily for Twelve Weeks in Adult Patients With Moderate-to-Severe Asthma Uncontrolled on Medium-High Dose ICS-LABA
Brief Title: Phase 2a Study to Assess the Efficacy and Safety of AZD4604 in Adult Patients With Moderate-to-Severe Asthma Uncontrolled on Medium-High Dose ICS-LABA
Acronym: AJAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8210C00003
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: asthma, Janus kinase inhibitor
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): AZD4604
  Interventions: Drug: AZD4604
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD4604 — AZD4604
  Arms: Arm 1
Other: Placebo — Placebo
  Arms: Arm 2

SUMMARY:
This is a Phase 2a, multicentre, randomised, placebo-controlled, double-blind, parallel-group study to evaluate the efficacy, safety and PK of AZD4604 administered BID using a dry-powder inhaler at one dose level over a 12-week Treatment period in adult participants with uncontrolled moderate-to-severe asthma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age inclusive, at the time of signing the informed consent.
2. Treated with medium-high dose ICS in combination with LABA at a stable dose for at least 28 days prior to Visit 1.

   Note: EU participants must be treated with high dose ICS in combination with LABA at a stable dose for at least 28 days prior to V1.
3. Documented history of ≥ 1 severe asthma exacerbation within 1 year prior to Visit 1.
4. Morning pre-BD FEV1 ≥ 40% predicted at Visit 1 and Visit 3.
5. Able to perform acceptable lung function testing for FEV1 according to ATS/ERS 2019 acceptability criteria.
6. Documented evidence of asthma in the 10 years up to or including Visit 1. A clinical diagnosis of asthma must be documented at least 12 months prior to Screening (Visit 1).
7. An ACQ-6 score ≥ 1.5 at Visit 1 and at Visit 3.

9. Body weight of ≥ 40 kg and body mass index of < 35 kg/m2. 10. Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. There are no restrictions on male participants or their female partners

At the end of the Run-in period (Visit 3), participants must fulfil the following additional criteria in order to be randomised into the study and enter the Treatment period:

1. Pre-BD FEV1 ≥ 40%.
2. A pre-BD/pre-IMP dose FEV1 at Visit 3 that has not increased or decreased by 20% or more from the pre-BD FEV1 recorded at Visit 1 and at Visit 2.
3. An ACQ-6 score of ≥ 1.5.
4. At least 80% compliance with usual asthma background medication during Run-in period (from Visit 2 to Visit 3) based on the daily asthma ePROs.
5. Minimum 80% compliance with daily eCOAs (electronic Clinical Outcome Assessments) during the 14 days preceding Visit 3.
6. For female of child bearing potential participants, a negative urine pregnancy test prior to administration of IMP.

Exclusion Criteria:

1. A severe asthma exacerbation within 8 weeks prior to randomisation.
2. History of herpes zoster reactivation.
3. Participants with a significant COVID-19 illness within 6 months of enrolment.
4. Clinically important pulmonary disease other than asthma.
5. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

   * affect the safety of the participant throughout the study,
   * influence the findings of the study or the interpretation, or
   * impede the participant's ability to complete the entire duration of study.
6. Any clinically significant cardiac or cerebrovascular disease.
7. History of venous thromboembolism.
8. Participants who, as judged by the investigator, have evidence of active TB, or latent TB without completion of an appropriate course of treatment or appropriate ongoing prophylactic treatment.
9. Participants with a recent history of, or who have a positive test for, infective hepatitis or unexplained jaundice, or participants who have been treated for HIV.
10. Current or prior history of alcohol or drug abuse (including marijuana and marijuana containing valid prescriptions), as judged by the investigator.
11. History of malignancy other than superficial basal cell carcinoma.
12. Treatment with systemic corticosteroid within 4 weeks (oral) or 8 weeks (intramuscular) before Visit 1.
13. Any immunosuppressive therapy within 12 weeks prior to Visit 1.
14. Treatment with marketed biologics within 6 months of Visit 1 or 5 half-lives, whichever is longer.
15. Inhaled corticosteroid plus fast-acting β2 agonist as a reliever is not allowed 15 days prior to Visit 1, during Screening/Run-in and throughout the Treatment period and preferably 1 week after the last dose of IMP.
16. Live, attenuated, or mRNA vaccines within 4 weeks of Visit 1.
17. Immunoglobulin or blood products within 4 weeks of Visit 1.
18. Any immunotherapy within 6 months of Visit 1, except for stable maintenance dose allergen-specific immunotherapy started at least 4 weeks prior to Visit 1 and expected to continue through to the end of the Follow-up period.
19. Concurrent enrolment in another interventional clinical study
20. Participant treated with any investigational drug within 4 months or 5 half-lives, whichever is longer, prior to Visit 1.
21. Participants with a known hypersensitivity to AZD4604 or any of the excipients of the product.
22. Abnormal findings identified on physical examination, ECG, or laboratory testing.
23. For female participants only - currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
24. Current smokers or participants with smoking history ≥ 10 pack-years.
25. Participants with a known long-term exposure to occupational asbestos, silica, radon, heavy metals, and polycyclic aromatic hydrocarbons.
26. Positive family history of primary lung cancer in first degree relatives (mother, father, sisters, brothers and children).
27. Positive urine cotinine test or exhaled carbon monoxide test at Visit 1 and at any timepoint throughout the study.
28. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
29. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
30. Donation of blood (≥ 450 mL) within 3 months or donation of plasma within 14 days before Visit 1.
31. Major surgery within 8 weeks prior to Visit 1, or planned inpatient surgery, major dental procedure or hospitalisation during Screening, Treatment, or Follow-up periods.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Time to first CompEx Asthma event | 12 weeks
  CompEx Asthma is a composite surrogate endpoint for exacerbations that captures: - acute worsening events based on a combination of events based on ePRO data (asthma symptoms and rescue medication use), PEF data, and severe asthma exacerbation events.

SECONDARY OUTCOMES:
Pre-BD FEV1 | 12 weeks
  Change from baseline in pre-bronchodilator forced expiratory volume in 1 second.
CAAT | 12 weeks
  Change from baseline in the Chronic Airways Assessment Test (CAAT). The CAAT is an 8-item patient-reported outcome measure developed to measure health status in patients with asthma and COPD.
ACQ-6 | 12 weeks
  Change from baseline in the Asthma Control Questionnaire 6 (ACQ-6). The ACQ-6 has 6 questions (regarding asthma symptoms and rescue bronchodilator use). Answering the questions results in a score out of 6. A Score of 0 indicates complete control and 6 reflects severely uncontrolled disease.
Average morning and average evening PEF | 12 weeks
  Change from baseline in 2-weekly average morning and evening Peak Expiratory Flow (PEF).
Daily asthma symptom score (total, daytime, and night-time) | 12 weeks
  Change from baseline in 2-weekly average Daily asthma symptom score. Asthma symptoms are assessed (0 to 3 scale) twice daily, once in the morning and once in the evening.
Time to first CompEx acute worsening event | 12 weeks
  Time to first CompEx Asthma acute worsening event.
CompEx event rate | 12 weeks
  The number of CompEx Asthma events recorded in the 12-week period.
CompEx acute worsening event rate | 12 weeks
  The number of CompEx Asthma acute worsening events recorded in the 12-week period.
FeNO | 12 weeks
  Change from baseline in FeNO at Week 4 and Week 12.
Cough | 12 weeks
  Change from baseline in cough severity at Week 4 and Week 12. This will be measured by Cough Severity Item Visual Analogue Scale, a 100-point linear scale marked with a horizontal or vertical line by the participant between the 2 extremes. Zero represents no cough while 100 represents worst cough imaginable.
PK | 12 weeks
  AZD4604 plasma concentration pre- and post-dose at Week 4, pre-dose at Week 12.

CONTACTS AND LOCATIONS:
Locations (110):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Newport Beach, California
  - Research Site, Sacramento, California
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hammond, Indiana
  - Research Site, New Bedford, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Saint Charles, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Union City, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Boerne, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Florida
  - Research Site, La Plata
  - Research Site, Ranelagh
- Brazil (6):
  - Research Site, Barretos
  - Research Site, Blumenau
  - Research Site, Campinas
  - Research Site, Porto Alegre
  - Research Site, São Bernardo do Campo
  - Research Site, São José do Rio Preto
- Research Site, Pazardzhik, Bulgaria
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, København Ø
  - Research Site, Vejle
- France (2):
  - Research Site, Lyon
  - Research Site, Strasbourg
- Germany (6):
  - Research Site, Berlin
  - Research Site, Cottbus
  - Research Site, Frankfurt am Main
  - Research Site, Koblenz
  - Research Site, Mainz
  - Research Site, Peine
- India (7):
  - Research Site, Ajmer
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Kozhikode
  - Research Site, New Delhi
- Malaysia (7):
  - Research Site, Kajang
  - Research Site, Kota Bharu
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Malacca
  - Research Site, Sarawak Miri
  - Research Site, Sungai Buloh
- Philippines (6):
  - Research Site, Dagupan
  - Research Site, Davao City
  - Research Site, Mabalacat
  - Research Site, Manadaluyong City
  - Research Site, Quezon City
  - Research Site, Roxas City
- South Africa (5):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Newton
  - Research Site, Observatory
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Palma de Mallorca
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Örebro
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
  - Research Site, Yunlin
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khlong Luang
  - Research Site, Khon Kaen
- United Kingdom (9):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Chesterfield
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Penzance
  - Research Site, Thetford
  - Research Site, Wellingborough
- Vietnam (7):
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh
  - Research Site, Hồ Chí Minh
  - Research Site, Huế